CLINICAL TRIAL: NCT03150979
Title: Effects of a Provision of a Cane on Locomotion and Social Participation of Individuals With Stroke: a Randomized Controlled Trial
Brief Title: Effects of a Provision of a Cane After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Luci Fuscaldi Teixeira-Salmela, Titular Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAPEMIG
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Stroke
Keywords: Stroke; Assistive devices; Gait; Rehabilitation; Clinical trial
MeSH Terms: conditions — Stroke | interventions — Canes

STUDY DESIGN:
Intervention Model Description: Prospective, single-blinded, randomized, clinical trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provision of a cane (Experimental): The experimental group will receive a single-point cane, with ergonomic handgrip, which will be individually adjusted to the participant's height. A physiotherapist will provide instructions on how to walk with the cane and the participants will practice for about 15 minutes or until they feel comfortable with the device. Then, they will take the cane home and will be instructed to use it all the time during locomotion. Weekly, they will receive a phone call, to ensure that they are using the cane and to clarify any doubts. A home visit may be conducted, if necessary.
  Interventions: Other: Provision of a cane
- Control (Other): The control group will be instructed to to perform stretching of the lower limb muscles daily and keep their daily activities, without the use of a cane. They will also receive weekly phone calls, to ensure similar level of attention to that of the the participants in the experimental group.
  Interventions: Other: Control

INTERVENTIONS:
Other: Provision of a cane — The participants will receive a single-point cane and will be instructed to use it all the time during locomotion. Weekly, they will receive a phone call, to ensure that they are using the cane and to clarify any doubts. A home visit may be conducted, if necessary.
  Arms: Provision of a cane
Other: Control — The control group will be instructed to to perform stretching of the lower limb muscles daily and keep their daily activities, without the use of a cane. They will also receive weekly phone calls, to ensure similar level of attention to that of the the participants in the experimental group.
  Arms: Control

SUMMARY:
Previous studies failed to determine the real effects of the provision of a walking cane after a stroke, mainly due to biases related to their methodological designs. In addition, there is no information on the carry-over effects of a cane to social participation. This study will test the hypothesis that the provision of a cane is effective in improving walking speed, step length, cadence, walking capacity, walking confidence, and participation of individuals with chronic stroke. For this prospective, single-blinded, randomized clinical trial, people after stroke will be randomly allocated into either experimental or control groups. The experimental group will receive a single-point cane, with ergonomic handgrip, which will be individually adjusted to the participant's height. A physiotherapist will provide instructions on how to walk with the cane and the participants will practice for about 15 minutes or until they feel comfortable with the device. Then, they will take the cane home and will be instructed to use it all the time during locomotion. Weekly, they will receive a phone call, to ensure that they are using the cane and to clarify any doubts. A home visit may be conducted, if necessary. The control group will be instructed to perform stretching of the lower limb muscles daily and keep their daily activities, without the use of a cane. To ensure the level of attention similar to that of the participants in the experimental group, the individuals in the control group will also receive weekly phone calls. At baseline (Week 0), post intervention (Week 4), and one month after the cessation (Week 8) of the interventions, researchers blinded to group allocations will collect all outcome measures.

DETAILED DESCRIPTION:
Rationale: Motor impairments after a stroke are disabling and interfere with the performance of daily activities, such as locomotion. Walking devices, such as a single cane, are usually prescribed to increase safety and improve gait ability. Previous studies failed to determine the real effects of the provision of a walking cane after a stroke, mainly due to biases related to their methodological designs. In addition, there is no information on the carry-over effects of a cane to social participation.

Aim: This study will test the hypothesis that the provision of a cane is effective in improving walking speed, step length, cadence, walking capacity, walking confidence, and participation of individuals with chronic stroke.

Design: For this prospective, single-blinded, randomized clinical trial, people after stroke will be randomly allocated into either experimental or control groups. The experimental group will receive a single-point cane, with ergonomic handgrip, which will be individually adjusted to the participant's height. A physiotherapist will provide instructions on how to walk with the cane and the participants will practice for about 15 minutes or until they feel comfortable with the device. Then, they will take the cane home and will be instructed to use it all the time during locomotion. Weekly, they will receive a phone call, to ensure that they are using the cane and to clarify any doubts. A home visit may be conducted, if necessary.

The control group will be instructed to perform stretching of the lower limb muscles daily and keep their daily activities, without the use of a cane. To ensure the level of attention similar to that of the participants in the experimental group, the individuals in the control group will also receive weekly phone calls. At baseline (Week 0), post intervention (Week 4), and one month after the cessation (Week 8) of the interventions, researchers blinded to group allocations will collect all outcome measures.

Study outcomes: walking speed, step length, cadence, walking capacity, walking confidence, and participation.

ELIGIBILITY:
Inclusion Criteria:

* People with stroke will be eligible if they are >6 months after the onset of their first stroke,
* >20 years of age,
* Able to walk at least 14 meters, independently, walk with a speed ≤0.8 m/s or less, and
* Are naïve to use any assistive device.

Exclusion Criteria:

* Individuals with cognitive impairments, double hemiparesis, or any other non-stroke related conditions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Walking speed | Baseline (week 0), after intervention (week 4) and one-month follow-up (week 8)
  Changes in walking speed, in m/s, assessed by the 10-m Walk Test.

SECONDARY OUTCOMES:
Walking step length | Baseline (week 0), after intervention (week 4) and one-month follow-up (week 8)
  Changes in walking step length, in meters, assessed by the 10-m Walk Test.
Walking cadence | Baseline (week 0), after intervention (week 4) and one-month follow-up (week 8)
  Changes in walking cadence, in step/minutes, assessed by the 10-m Walk Test.
Walking capacity | Baseline (week 0), after intervention (week 4) and one-month follow-up (week 8)
  Changes in walking capacity, in meters, assessed by the 6-min Walk Test.
Walking confidence | Baseline (week 0), after intervention (week 4) and one-month follow-up (week 8)
  Changes in walking confidence, reported as scores ranging from 10 to 100, assessed by the Modified Gait Efficacy Scale.
Social Participation | Baseline (week 0), after intervention (week 4) and one-month follow-up (week 8)
  Changes in social Participation, assessed by the Stroke Impact Scale (social participation sub-section).

CONTACTS AND LOCATIONS:
Overall Officials: Luci F Teixeira-Salmela, Ph.D., Principal Investigator — Federal University of Minas Gerais
Locations (2):
- Brazil (2):
  - Department of Physical Therapy, Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - NeuroGroup Laboratory, Belo Horizonte, Minas Gerais

IPD SHARING:
Plan to Share IPD: No